CLINICAL TRIAL: NCT00822133
Title: Percutaneous Ketamine Versus Lidocaine or Placebo, for Post-Surgery Analgesia, in Patients Undergoing Laparoscopic Partial Lung Resection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: AA Weinbroum, MD, Tel Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0250-08-TLV
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Last update posted 2009-01-14 (Estimated); Status verified 2009-01

CONDITIONS: Postoperative Pain
Keywords: ketamine; preemption; postoperative; pain; safety
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Lidocaine; Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- lodocaine (Active Comparator): lidocaine 5% cream will be put on the skin
  Interventions: Drug: lidocaine
- ketamine (Experimental): ketamine 5% will be put on the skin
  Interventions: Drug: ketamine
- placebo (Placebo Comparator): non-active cream will be put on the skin
  Interventions: Drug: non-active drug cream

INTERVENTIONS:
Drug: lidocaine — lidocaine 5%
  Arms: lodocaine
Drug: ketamine — ketamine cream
  Arms: ketamine
Drug: non-active drug cream — will be put on the skin
  Arms: placebo

SUMMARY:
Since VAT bears with it severe postopearive pain, and since ketamine has been shown to be an optimal analgesics adjuvant for postoperative pain, we wish to assess to effects of ketamie vs. lidocaine if put on the skin in the sites where scopes are interset into the chest for thoracoscopy.

DETAILED DESCRIPTION:
Ketamine hydrochlorid is a general anesthetic that is also used as short term sedative. Ketamine has an antagonistic effect on the central spinal N-Methyl-D-Aspartate (NMDA) receptors, the latter modulating pain stimuli generated peripherally on their way to central pain centers.

Ketamine has been used recently pre-operatively rather than post-operatively. Our recent experience with pre-operative use of ketamine has not been analyzed yet by Tel Aviv Medical Center's researchers. However, there is some experience with topical dermal, epidural, intra-articular and oral usage of ketamine.

As far as we no, there are no reports on patients' subjective feeling when ketamine was given pre-operatively for postoperative acute pain in patients undergoing partial lung resections. The possible influence of such an effect on the patient's well-being and the patient's family feelings and reactions were neither explored.

The goal of the study is to examine the possibility that if ketamine is administered in the pre-operative period, as a topical ointment, this will induce changes in the patient's sensation of pain, his own satisfaction, and possibly his family's satisfaction as well. The basis of this contention is that by administering less morphine (which is given to the patient in the immediate post-operative period through PCA [Patient-Controlled Analgesia]), with or without changes in pain, might have positive effects on the patient's well being and his family's. This issue will be assessed by a verbal questionnaire and based and on a visual analog scale (VAS).

Three groups of 20 patients each will be enrolled in the study. The first group will receive a placebo topical paste which will be produced by the hospital pharmacy. The second group will be given Lignocain paste, and the third group will get ketamine topical paste, prepared by the pharmacy as well. The study will be double blind and randomized. All patients will be treated with morphine postoperatively, as mentioned above.

It is anticipated that the amounts of morphine that will be used by the patients postoperatively by patients treated by ketamine will be reduced as compared to the other groups. This might increase the patient's and family's satisfaction rates, regardless of the decrease in the subjective pain ratings.

The importance of this study is that if the contention that is at the basis of this study is proven true, similar surgical groups of patients will benefit from the addition of topical ketamine administration to the habitual morphine-used postoperative only analgesia. By doing so, complications that stem from high doses of morphine will diminish, thus maintain hemodynamic stability and benefiting from the advantages of a patient being awake, cooperative and able to feedback the medical personnel in real time about his condition. Cooperation and satisfaction of the patient and family could be the end result of this process. Finally, it is assumed that under such conditions the number of complications in the postoperative period will minimize as well.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing VAT

Exclusion Criteria:

* emergency patients, open thoracotomy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-06 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
reduce postoeprative pain | up to 3 months

SECONDARY OUTCOMES:
overall patient satisfaction | up to 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky Medical center, Tel Aviv, Israel